CLINICAL TRIAL: NCT00321945
Title: A Retrospective Analysis of the Use of ACE-inhibitors and Angiotensin Receptor Blockers on Post-Operative Atrial Fibrillation
Brief Title: A Retrospective Analysis of the Use of ACE-inhibitors and Angiotensin Receptor Blockers
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., Principal Investigator, Emory University
Other Study IDs: IRB00002174
Record Dates: First submitted 2006-05-01; First posted 2006-05-04 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Angiotensin Converting Enzyme Inhibitor; Angiotensin Receptor Blocker
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ACE-Inhibitors and Angiotensin Receptor Blockers — Retrospective study - no intervention as part of study.

SUMMARY:
It is well known that atrial fibrillation (AF) and atrial flutter occur frequently after most types of cardiac surgeries.(1-4) Postoperative AF is associated with significant morbidity, longer hospital stay, and higher related costs. Currently, it is common procedure to premedicate patients with antiarrhythmic drugs for elective cardiac surgeries. Treatments such as beta blockers, Amiodarone, and electrical pacing are used to help prevent the morbidity associated with pot-operative AF.(5)

Renin-angiotensin system (RAS) activation may contribute to AF. Several clinical trials have suggested that inhibitors of this system may reduce the incidence of AF.(6-12) Patients with AF are known to have increased levels of angiotensin converting enzyme (ACE) and some types of angiotensin receptors.(13-15) Data from animal studies performed by our group suggest that cardiac ACE overexpression may lead to arrhythmic ion channel changes.(16;17) Although not studied in this group yet, it would be reasonable to conclude that the use of ACE inhibitors and angiotensin receptor blockers (ARBs) would decrease the incidence of AF in post-operative patients, too

DETAILED DESCRIPTION:
2.0 Objectives

Based on the discussion above, we hypothesize that patients premedicated on ACE Inhibitors and ARBs will have a decreased incidence of post-operative AF or atrial flutter. This study will be a retrospective cohort analysis of all patients that underwent elective cardiac surgeries between 2000-2005 at Emory University Hospital, Crawford Long Hospital, or the Atlanta Veterans Affairs Medical Center to evaluate the relationship of pre-operative ACE inhibitor or ARB use to the incidence of post-operative atrial arrhythmias.. This study is undertaken in preparation for a funding proposal for a prospective trial.

3.0 Patient Selection 3.1 Eligibility criteria:

1. All patients that patients who underwent elective cardiac surgery in the Emory University Hospital, Crawford Long Hospital, or the VA Medical Center between 2000-2005.

3.2 Ineligibility criteria:

1. Emergent operations.
2. The presence of AF or atrial flutter at the time of surgery.
3. Patients without adequate documentation of atrial rhythm following surgery.
4. New York Heart Association (NYHA) class IV heart failure at the time of surgery.
5. Hyperthyroidism
6. Implanted devices for designed for active management of atrial arrhythmias by pacing or defibrillation
7. Known illicit drug use
8. Known ethanol abuse
9. Electrophysiological ablation for atrial tachycardia within 6 months of the operation.

4.0 Registration and randomization: none

5.0 Therapy: none

6.0 Pathology: none

7.0 Patient assessment: none

8.0 Data collection: Data will be collected from review of the patient's hospital charts, from telemetry recordings, and ECGs to document the presence or absence of AF or atrial flutter during the hospital admission for cardiac surgery. The presence or absence of atrial fibrillation will be diagnosed on the basis of an electrocardiographic recording and confirmed by a cardiologist. Demographic data collected will include: age, race, sex, body mass index, blood pressure, NYHA classification, Killip classification, and the history of previous myocardial infarction, hypertension, diabetes, smoking, alcohol use, antiarrhythmic drug use, presence and type of pacemaker if any, history of AF or atrial flutter, previous cardiovascular events, type of operation, and length of operation. Patients enrolled in this study will be given unique study numbers. No follow up data will be required from patients.

9.0 Statistical considerations: This study design is a retrospective chart review of a cohort of patients undergoing cardiac surgery to determine if there is an association between pre-operative ARB or ACE inhibitor use and the incidence of post-operative atrial fibrillation or atrial flutter. The null hypothesis is that there is no association between the preoperative use of ACE Inhibitors and ARBs and postoperative AF and atrial flutter. Within the cohort, those patients with AF or atrial flutter will be compared to those without these atrial arrhythmias in the post-operative period. Baseline data for the two groups will be expressed as mean ± standard deviation for continuous variables, and frequencies for categorical variables. Differences in baseline characteristics between the groups will be examined by use of Fisher exact and Mann-Whitney tests for categorical and continuous variables, respectively. Quantification of any association between pre-operative ACE Inhibitors and ARBs and the presence of atrial fibrillation will modeled by logistical regression analysis after adjusting for other variables that may affect arrhythmia frequency.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent elective cardiac surgery in the Emory University Hospital, Crawford Long Hospital, or the VA Medical Center between 2000-2005.

Exclusion Criteria:

* Emergent operations.
* The presence of AF or atrial flutter at the time of surgery.
* Patients without adequate documentation of atrial rhythm following surgery.
* NYHA class IV heart failure at the time of surgery.
* Hyperthyroidism
* Implanted devices for designed for active management of atrial arrhythmias by pacing or defibrillation
* Known illicit drug use
* Known ethanol abuse
* Electrophysiological ablation for atrial tachycardia within 6 months of the operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, 18 years or older up to and including 65 years of age, who underwent elective cardiac surgery in the Emory University Hospital, Crawford Long Hospital, or the VA Medical Center between 2000-2005.
Sampling Method: Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the relationship of pre-operative ACE inhibitor or ARB use to the incidence of post-operative atrial arrhythmias. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Dudley, Jr., MD, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Crawford Long Hospital, Atlanta, Georgia
  - Veterans Administration Medical Center, Decatur, Georgia